CLINICAL TRIAL: NCT03672617
Title: Validation of a Patient-reported Outcome (PRO) Measure That Assesses Reasons for Non-adherence to Growth Hormone Therapy (GHT)
Brief Title: Validation of a Questionnaire That Identifies the Reasons for Non-adherence to Existing Growth Hormone Therapy
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: GH-4415; U1111-1210-1036 (Other: World Health Organization (WHO))
Record Dates: First submitted 2018-09-07; First posted 2018-09-14 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Growth Hormone Deficiency in Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children and adolescents: Children and adolescents, who administer growth hormone (GH) themselves (self-injections) will be asked to complete the questionnaire.
  Interventions: Other: No treatment given
- Parents/legal guardians: Parents/legal guardians who administer the GH to their child will be asked to complete the questionnaire.
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — No treatment is given to study participants. Only evaluation of a questionnaire assessing reasons for non-adherence to growth hormone therapy (GHT) and to determine its validity and reliability.
  The preliminary working title of the questionnaire GHCQ used in the outcome measures was renamed for simplicity reasons into BAR-GHT (abbreviation for barriers to growth hormone therapy) after study completion.

SUMMARY:
The aim of the study is to examine the suitability, the so-called validation, of a questionnaire, with which one can grasp the reasons why injections of growth hormones are omitted by patients ("non-adherence"). Participants are treated with growth hormone and are therefore eligible to take part in the study. Study doctor will ask participants to answer questionnaires. two times within 14 days. The first time participants answer during the routine visit to the practice / clinic and the second time at home. There are no risks associated with participating in the study as it does not affect participant's medical treatment.

ELIGIBILITY:
Inclusion Criteria: - Children/adolescents, male or female, aged 8 to 18 years who self-inject GH as well as their parents/legal guardians or Parents/Legal guardians who administer GH to a child/adolescent, male or female, from birth to 18 years - The child/adolescent is on prescribed daily GHT due to idiopathic growth hormone deficiency (GHD), multiple pituitary hormone deficiency (MPHD/organic GHD), small for gestational age (SGA) or Turner syndrome (TS) for at least 6 months before screening visit - Signed informed consent obtained by parent/legal guardian and child/adolescent before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol) Exclusion Criteria: - Mental incapacity, unwillingness or language barrier of participant precluding adequate understanding or cooperation - Previous participation of participant in this study. Participation is defined as having given informed consent in this study - Treatment of child/adolescent with any investigational drug within 30 days prior to enrolment into the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Three hundred (300) participants at about 30 sites for paediatric endocrinology in Germany will be included in this validation study.
Sampling Method: Non-Probability Sample
Enrollment: 321 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-04-25 (Actual)

PRIMARY OUTCOMES:
Validity of the Growth Hormone Compliance Questionnaire child/adolescent version (GHCQ-CA) | Day 1
  The GHCQ-CA is a patient-reported outcome measure designed to assess reasons for non-adherence to growth hormone therapy in children/adolescents from the child's/adolescent's perspective. The GHCQ-CA currently has 34 items. All GHCQ-CA questions are answered on a 5-point Likert scale from 'Never' to 'Always'.
Validity of the GHCQ-CA | Day 14
  The GHCQ-CA is a patient-reported outcome measure designed to assess reasons for non-adherence to growth hormone therapy in children/adolescents from the child's/adolescent's perspective. The GHCQ-CA currently has 34 items. All GHCQ-CA questions are answered on a 5-point Likert scale from 'Never' to 'Always'.
Reliability of the GHCQ-CA | Day 1
  The GHCQ-CA is a patient-reported outcome measure designed to assess reasons for non-adherence to growth hormone therapy in children/adolescents from the child's/adolescent's perspective. The GHCQ-CA currently has 34 items. All GHCQ-CA questions are answered on a 5-point Likert scale from 'Never' to 'Always'.
Reliability of the GHCQ-CA | Day 14
  The GHCQ-CA is a patient-reported outcome measure designed to assess reasons for non-adherence to growth hormone therapy in children/adolescents from the child's/adolescent's perspective. The GHCQ-CA currently has 34 items. All GHCQ-CA questions are answered on a 5-point Likert scale from 'Never' to 'Always'.
Validity of the Growth Hormone Compliance Questionnaire parent version (GHCQ-P) | Day 1
  The GHCQ-P is a patient-reported outcome measure designed to assess reasons for non-adherence to growth hormone therapy in children/adolescents from the parents'/legal guardian's perspective. The GHCQ-P currently has 50 items. All GHCQ-P questions are answered on a 5-point Likert scale from 'Never' to 'Always'.
Validity of the GHCQ-P | Day 14
  The GHCQ-P is a patient-reported outcome measure designed to assess reasons for non-adherence to growth hormone therapy in children/adolescents from the parents'/legal guardian's perspective. The GHCQ-P currently has 50 items. All GHCQ-P questions are answered on a 5-point Likert scale from 'Never' to 'Always'.
Reliability of the GHCQ-P | Day 1
  The GHCQ-P is a patient-reported outcome measure designed to assess reasons for non-adherence to growth hormone therapy in children/adolescents from the parents'/legal guardian's perspective. The GHCQ-P currently has 50 items. All GHCQ-P questions are answered on a 5-point Likert scale from 'Never' to 'Always'.
Reliability of the GHCQ-P | Day 14
  The GHCQ-P is a patient-reported outcome measure designed to assess reasons for non-adherence to growth hormone therapy in children/adolescents from the parents'/legal guardian's perspective. The GHCQ-P currently has 50 items. All GHCQ-P questions are answered on a 5-point Likert scale from 'Never' to 'Always'.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Mainz, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com/sharing-results

REFERENCES:
- [Derived] de Zwaan M, Fischer-Jacobs J, Wabitsch M, Reinehr T, Meckes-Ferber S, Crosby RD. Development and Psychometric Evaluation of an Instrument Assessing Barriers to Growth Hormone Treatment (BAR-GHT). Front Endocrinol (Lausanne). 2020 Feb 25;11:84. doi: 10.3389/fendo.2020.00084. eCollection 2020. PMID 32158432